CLINICAL TRIAL: NCT00465348
Title: The Antioxidant Effect of Routine Vascular Therapy for Normal Tension Glaucoma Patients
Status: Withdrawn | Type: Observational
Why Stopped: investigator withdrew
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 085-Mom-2007
Record Dates: First submitted 2007-04-24; First posted 2007-04-25 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Primary Open Angle Glaucoma
Keywords: normal tension glaucoma; vascular dysregulation
MeSH Terms: conditions — Glaucoma, Open-Angle; Low Tension Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
To quantify oxidative stress in circulating leukocytes of normal tension glaucoma patients, prior to and one month after routine vascular therapy.

DETAILED DESCRIPTION:
There are two accepted medical modalities for glaucoma treatment. The first, is a local application of an intraocular pressure (IOP) lowering drug. The second, is the application of systemic drugs to improve vascular regulation. In the present study we would like to investigate whether this systemic form of treatment, in addition to improving blood flow, also reduces systemic oxidative stress.

Vascular dysregulation is one of the major risk factors for glaucoma, in particular for normal tension glaucoma (NTG). In glaucoma patients blood flow is, on average, reduced not only in the eye but also in various other organs of the body, for example in the fingers. Such a systemic dysregulation leads to disturbed autoregulation and thereby to an unstable oxygen supply in the eye.This, in turn, leads to the formation of reactive oxygen species (ROS). These ROS are capable of damaging cells such as white blood cells; this damage, however, is reversible as nature has provided us with mechanisms to repair this damage. This reversible damage brought about by ROS, which is constantly being repaired in our body, is an indication for oxidative stress. Oxidative stress plays an important role in the pathogenesis of glaucoma.

The indications for oxidative stress can be quantified in our laboratory by the method of comet assay also known as single cell gel electrophoresis.

ELIGIBILITY:
Inclusion Criteria:

For NTG patients:

* A mean untreated intraocular pressure consistently equal to or below 21mmHg or median intraocular pressure equal to or below 20mmHg on diurnal testing (at least three measurements) with no single measurement greater than 24mmHg
* Open drainage angles on gonioscopy
* Typical optic disc damage with glaucomatous cupping and thinning of neuroretinal rim
* Visual field defect congruent to glaucomatous disc alteration
* No other pathological findings upon slit-lamp examination and indirect fundoscopy
* Vasospastic propensity will be assumed if a clear history of frequent cold hands (answering yes to the questions:" Do you always have cold hands, even during the summer time?" and "Do other people tell you that you have cold hands?") is reported.

For healthy subjects:

* An intraocular pressure < 20 mmHg
* No history of ocular or systemic disease
* No history of chronic or current systemic or topical medication, or of drug or alcohol abuse
* Normal blood pressure (100-140/60-90mm Hg)
* Best corrected visual acuity above 20/32 in both eyes
* No pathological findings upon slit-lamp examination and indirect fundoscopy

Exclusion Criteria:

EXCLUSION CRITERIA:

* Iridocorneal angle extremely narrow with complete or partial closure as determined by gonioscopy
* Pigmentary dispersion or pseudoexfoliation
* Evidence for any secondary cause for a glaucomatous optic neuropathy (trauma, steroids, uveitis)
* History of chronic or recurrent severe inflammatory eye disease (eg. scleritis, uveitis) or clinically significant or progressive retinal disease (eg. diabetic retinopathy)
* History of ocular trauma or intraocular surgery within the past 6 months
* History of systemic infection or inflammation within the past 3 months
* Need for any concomitant medications that may interfere with the evaluation of leukocytes (eg: steroids, immunosuppressives)
* Patients with a significant history and /or active alcohol or drug abuse (significant is defined as that which may influence results of the study)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary open-angle glaucoma patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Selim Orgül, MD, Study Director — University Hospital Basel, Eye Clinic

REFERENCES:
- [Background] Moenkemann H, Flammer J, Wunderlich K, Breipohl W, Schild HH, Golubnitschaja O. Increased DNA breaks and up-regulation of both G(1) and G(2) checkpoint genes p21(WAF1/CIP1) and 14-3-3 sigma in circulating leukocytes of glaucoma patients and vasospastic individuals. Amino Acids. 2005 Mar;28(2):199-205. doi: 10.1007/s00726-005-0169-x. Epub 2005 Jan 23. PMID 15723242